CLINICAL TRIAL: NCT03661645
Title: Post-operative Methylprednisolone Taper Course for Orthopedic Surgery
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Michael Gottschalk, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00104310
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Orthopedic Surgeries
Keywords: Glucocorticoids(GS); injection
MeSH Terms: interventions — Dexamethasone; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized Controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methylprednisolone Treated Group (Active Comparator): Subjects in this group will receive single intraoperative course of 10 mg IV dexamethasone & 6 day oral methylprednisolone taper that is 10 mg Intravenous IV dexamethasone and 6 day oral methylprednisolone taper course
  Interventions: Drug: 10 mg IV dexamethasone & 6 day oral methylprednisolone taper
- Control Group (Other): Subjects in this group will receive single intraoperative dose of 10 mg IV dexamethasone; that is 10 mg Intravenous (IV) dexamethasone
  Interventions: Other: 10 mg IV dexamethasone

INTERVENTIONS:
Drug: 10 mg IV dexamethasone & 6 day oral methylprednisolone taper — Drug: 6-day oral methylprednisolone (glucocorticoid) taper course The oral methylprednisolone taper course will begin on the day of surgery and will include 24mg on day 1, 20mg on day 2, 16mg on day 3, 12mg on day 4, 8mg on day 5, and 4mg on day.
  Drug:10 mg intravenous (IV) dexamethasone
  Other Names: Medrol, Depo-Medrol, Solu-Medrol, A-Methapred; Decadron, Dexasone, Diodex, Hexadrol, Maxidex
  Arms: Methylprednisolone Treated Group
Other: 10 mg IV dexamethasone — Drug:10 mg intravenous (IV) dexamethasone
  Other Names: Decadron, Dexasone, Diodex, Hexadrol, Maxidex
  Arms: Control Group

SUMMARY:
The clinical trial is a prospective randomized control trial of a group of patients undergoing surgical management of common orthopedic pathologies including fractures of the upper extremity and shoulder arthroplasty; arthritis surgeries (ex. carpometacarpal arthroplasty), release of compressive neuropathies (ex. carpal tunnel surgery), tendon procedures (ex. tendon repair), patients undergoing total hip arthroplasty for osteoarthritis of the hip or total knee arthroplasty for osteoarthritis of the knee.

Patients will be assigned randomly to one of two treatment arms: (1) single intraoperative dose of 10 mg intravenous dexamethasone (control group, IV dexamethasone is standard of care) or (2) single intraoperative dose of 10 mg intravenous dexamethasone followed with a 6-day oral methylprednisolone taper course (Active Group).

The purpose of this study is to study the efficacy of a post-operative course of glucocorticoids (GCs like Methylprednisolone) on pain, nausea and range of motion after surgical management of common orthopedic upper extremity pathologies, including fractures of the upper extremity and shoulder arthroplasty and patients undergoing total hip arthroplasty for osteoarthritis of the hip or total knee arthroplasty for osteoarthritis of the knee.

DETAILED DESCRIPTION:
Reducing pain and improving function is of great importance in the immediate period after surgery. Many orthopaedic procedures result in fluid build-up around the surgical site which results in pain and decreased healing. Glucocorticoids are drugs that block the inflammatory process which can decrease this pain and fluid build-up. Furthermore, glucocorticoids are safe if given in low doses and for a short period of time. To help address this gap, the study intend to give patients glucocorticoids after various upper extremity orthopedic procedures; total hip arthroplasty for osteoarthritis of the hip or total knee arthroplasty for osteoarthritis of the knee, assessing their pain and range of motion post-operatively. The study hypothesize that glucocorticoids will result in less inflammation around the surgical site, leading to pain relief, greater healing ability, and improvements in range of motion of the injured joint.

The study aims to enroll 500 subjects that are assigned randomly to one of two treatment arms: (1) single intraoperative dose of 10 mg intravenous dexamethasone (control group), IV dexamethasone is standard of care) or (2) single intraoperative dose of 10 mg intravenous dexamethasone followed with a 6-day oral methylprednisolone taper course (active group). Subjects will be followed up in clinic 2, 6, and 12 weeks postoperatively that is a standard of care for upper extremity fractures, shoulder arthroplasty, total hip arthroplasty for osteoarthritis of the hip or total knee arthroplasty for osteoarthritis of the knee

ELIGIBILITY:
Inclusion Criteria:

* Patients of Emory Hand Surgeons undergoing surgery for an upper extremity fracture who are willing to participate in the study will be included in the study (Including American Orthopedic(AO) and American Orthopaedic Trauma Association (OTA) AO/OTA Classification 1, 2, and 7 +/- Type A, B, C).
* Patients of Emory Hand Surgeons undergoing Total Shoulder Arthroplasty or Reverse Shoulder Arthroplasty who are willing to participate in the study will be included in the study (Walsh Classification A-D).
* Patients of Emory Hand Surgeons undergoing surgery for upper extremity arthritis (ex. carpometacarpal arthroplasty)
* Patients of Emory Hand Surgeons undergoing release for upper extremity compressive neuropathies (ex. carpal tunnel surgery)
* Patients of Emory Hand Surgeons undergoing procedures for upper extremity tendon pathologies (ex. tendon repair)
* Patients undergoing total hip arthroplasty for osteoarthritis of the hip
* Patients undergoing total knee arthroplasty for osteoarthritis of the knee
* Between the ages of 18 years and 95 years.
* Patients willing and able to provide written and informed consent

Exclusion Criteria:

* Patients with concurrent and significant injuries to other bones or organs.
* Patients with local infections.
* Patients who are minors, vulnerable subjects, or who are not willing to consent to participate in the study.
* History of alcohol or medical abuse, allergies to glucocorticoids, daily use of glucocorticoids or chronic opioid use prior to the injury (morphine, fentanyl, hydromorphone, ketobemidone, methadone, nico morphine, oxycodone, and meperidine), history of severe heart disease ( New York Heart Association (NYHA 2)), renal failure, or liver dysfunction, active peptic ulcer disease, diabetic neuropathy, rheumatoid arthritis, and neurological or psychiatric diseases, potentially influencing pain perception.
* Women who are pregnant
* Patients with pre-existing immune suppression, where further immune suppression with GCs could warrant unwarranted or unneeded risk.
* Subjects who, in the opinion of the investigator, may be non-compliant with study schedules or procedures.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-09-07 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change in post-operative pain scores using numeric verbal analogue scores (VAS-Pain) during follow up in the methylprednisolone treated group compared to the control group | Post Operative day (1-15), 2 weeks, 6 weeks, 12 weeks, and 1 year postoperatively
  Pain assessment will be assessed before performing the injection, at the time of injection, and at each subsequent follow up visit using the Visual Analog Pain Scale (VAS-pain). The pain VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. Pain will be assessed at rest and active movement of the affected joint. Cut points for VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm). Normative values are not available.
Change in post-operative nausea scores using numeric verbal analogue scores (VAS-Nausea) during follow up in the methylprednisolone treated group compared to the control group | Post Operative day (1-15), 2 weeks, 6 weeks, 12 weeks, and 1 year postoperatively
  The (VAS-Nausea) questionnaire is self-completed by the subject. Subject is asked to place a line perpendicular to the VAS line at the point that represents their nausea severity.Subjects will rate their nausea severity on a 10-cm visual analog scale. The scale is ranked from 0 (least severe) to 10 (most severe).
Change in Range of Motion (ROM) prior to surgery and during follow up in the methylprednisolone treated group compared to the control group | Pre operatively, 2 weeks, 6 weeks, 12 weeks, and 1 year postoperatively
  ROM assessment will take place at each clinic follow up with a hand-held goniometer. . This will be done by assessing the total flexion-extension arc of the wrist, elbow, shoulder, knee, or hip; the total pronation-supination arc at the wrist; and the adduction-abduction arc of the wrist, shoulder, and hip. ROM will be assessed on the contralateral side prior to surgery.
Change in postoperative Quick Disabilities of Arm, Shoulder and Hand (QuickDASH) scores during follow up in the methylprednisolone treated group compared to the control group among subjects that underwent surgical management for upper extremity injuries | 2 weeks, 6 weeks, 12 weeks, and 1 year postoperatively
  The domains explored by the Quick DASH are: (1) physical arm, shoulder or hand activity problems (6 items); (2) severity of pain and tingling (2 items); (3) social activities, work, and sleep (3 items). Each item has five response options, ranging from 1, ''no difficulty or no symptom,'' to 5, ''unable to perform activity or very severe symptom.'' If at least 10 of the 11 items are completed, a score ranging from 0 (no disability) to 100 (most severe disability) can be calculated [(sum of n responses/n) - 1] x 25.the effect size and the percentage of patients reaching Minimal Clinical Important Improvement was determined.
Change in postoperative American Shoulder and Elbow Surgeons Shoulder Score (ASES) during follow up in the methylprednisolone treated group compared to the control group among subjects that underwent surgical management for upper extremity injuries | 2 weeks, 6 weeks, 12 weeks, and 1 year postoperatively
  The American Shoulder and Elbow Surgeons Shoulder Score (ASES) is a mixed outcome reporting measure, applicable for use in all patients with shoulder pathology for the assessment of shoulder function. The ASES questionnaire is composed of 17 questions. The questions focus on joint pain, instability, and activities of daily living. It is a 100 point scale (Pain scale= 50 points, 10 activities of daily living = 50 points).Score range: Pain subscale 0-50 ASES points; function/disability subscale 0-50 ASES points. Total score 0-100 ASES points (0 = worse pain and functional loss/disability).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gottschalk, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Clinic A, Clifton Road Clinic, Atlanta, Georgia
  - 21 Ortho Lane, Atlanta, Georgia
  - Emory Healthcare Orthopaedics and Spine Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wagner ER, Hussain ZB, Karzon AL, Cooke HL, Toston RJ, Hurt JT, Dawes AM, Gottschalk MB. Methylprednisolone taper is an effective addition to multimodal pain regimens after total shoulder arthroplasty: results of a randomized controlled trial: 2022 Neer Award winner. J Shoulder Elbow Surg. 2024 May;33(5):985-993. doi: 10.1016/j.jse.2023.12.016. Epub 2024 Feb 4. PMID 38316236